CLINICAL TRIAL: NCT03725488
Title: The Impact of Background Music in Reducing Stress in Preclinical Dental Labs
Status: Completed | Type: Observational
Sponsor: Ajman University (Other)
Responsible Party: Principal Investigator, sudhir rama varma, ASSISTANT PROFESSOR, Ajman University
Other Study IDs: RDF-2015/16-01
Record Dates: First submitted 2018-10-10; First posted 2018-10-31 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Stress-related Problem
Keywords: Dental labs; genre; music; perceived stress scale; stress
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Active: Evaluate stress among dental students by Questionnaire
  Interventions: Other: Questionnaire
- the present level of stress, comfort zone & coping with stress: Evaluate how stress was coped, the coping mechanisms used through Questionnaire
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — students were involved in the pre-clinical prosthodontic lab. Participation in these labs were mandatory and it involved crown and bridge preparations on typodont models. There were 2 sessions of these labs per week, one for each gender. Each session lasted for 3 hours.
  The study was conducted in 2 phases. At the beginning of the first phase of the study, the labs were conducted without any BM for 4 weeks. PSS(perceived stress scale), a standardized and validated, self-reporting international test was used for measuring the level of psychological stress were administered to all participants.

SUMMARY:
This study was designed to evaluate students' level of stress and impact of background music on their efficiency of work, performance and learning ability during pre-clinical lab.

DETAILED DESCRIPTION:
The reported high level of stress among dental students and its consequences, considering the known benefits of background music. This study was designed to evaluate students' level of stress and impact of background music on their efficiency of work, performance and learning ability during pre-clinical lab.

METHODOLOGY: In this cross-sectional questionnaire study, 61 preclinical students from the college of dentistry, Ajman university-Fujairah campus who met the defined inclusion criteria participated.

After a semester of the normal lab without BM (Background Music), various genres of BM were introduced in the lab. Psychological stress assessment was done using P.S.S (Perceived Stress Scale).Students were asked to fill up a written feedback questionnaire at the end of six weeks of BM. Descriptive statistics and Chi-square test were used in order to study the statistical relationships among groups.

ELIGIBILITY:
Inclusion Criteria:

* Students were not taking any
* medication for anxiety
* did not suffer from depression
* did not have any systemic illness;
* and they had no aversion towards music.

Exclusion Criteria:

* Students who were taking
* medication for anxiety
* had depression
* had systemic illness
* they had aversion towards music

Ages: 18 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population were both male and female students aged between 18-23 yrs who were students of Ajman University dental campus,they are attending preclinical dental labs and belong to the 2nd and third year of the dentistry program
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-02-24 (Actual); Primary Completion 2016-07-25 (Actual); Study Completion 2016-08-20 (Actual)

PRIMARY OUTCOMES:
coping mechanisms practiced by pre-clinical dental students to cope up stress. | From baseline to 5 months
  How students cope with the stress they experience by answering a questionnaire
PSS ((perceived stress scale) internationally used psychological scale for measuring the level of stress, it measures how stressful are the situations in one's life.) | From baseline to 5 months
  It consist of ten questions, each question has five answers arranged from zero to four. Each number has a point which reveals the level of stress for each question. Points were calculated according to the calculation system of the scale.
PSS scale range from 0-4,with 0-no stress,1-mild stress,3-moderate stress and 4-severe stress | From baseline to 5 months
  The students were graded on their response to the questionnaire

SECONDARY OUTCOMES:
Feedback of music of male and female pre-clinical dental students. | From baseline to 5 months
  What type of music students feel more relaxed while working in dental labs by answering certain questions in the form of questionnaire
PSS scale range from 0-4,with 0-no stress,1-mild stress,3-moderate stress and 4-severe | From Baseline to 5 months
  What type of music students feel more relaxed while working in dental labs by asking certain questions in a questionnaire
  a measurement tool in the form of questionnaire

IPD SHARING:
Plan to Share IPD: Yes
Results of the study,also methodology
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2 months